CLINICAL TRIAL: NCT06858943
Title: Can Tendon Autograft Function As a Meniscal Transplant
Acronym: DR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed hussein khalil, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N 207-2024
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Meniscectomy
Keywords: Meniscus ; Peroneus longus autograft

STUDY DESIGN:
Intervention Model Description: case series of 25 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arthroscopic meniscus reconstruction using a tendon autograft (Experimental): arthroscopic meniscus reconstruction using a tendon autograft
  Interventions: Procedure: arthroscopic meniscus reconstruction using a tendon autograft

INTERVENTIONS:
Procedure: arthroscopic meniscus reconstruction using a tendon autograft — arthroscopic meniscus reconstruction using a tendon autograft

SUMMARY:
Purpose: To evaluate the functional outcomes after using peroneus longus (PL) tendon autograft as meniscal transplantation in patients with knee joint line pain exaggerated with weight bearing following prior total or subtotal meniscectomy.

DETAILED DESCRIPTION:
This research design is a single center prospective study carried out at a tertiary trauma center hospital between May 2022 and December 2022. This research had ethical Committee Approval which was granted by the Ethics Committee of Cairo University (Institutional Review Board (IRB) number N 207-2024). All patients signed an informed consent before joining this study. This study included 25 patients, with previous history of subtotal or total meniscectomy medially or laterally, who underwent meniscus transplantation using PL tendon autograft.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients with a history of prior subtotal or total (medial or lateral meniscus) meniscectomy.
* Post meniscectomy symptoms (medial or lateral knee joint line pain exaggerated with weight bearing).

Exclusion Criteria:

* Multi-ligamentous knee injuries.
* Skeletally immature patients.
* Significant osteoarthritic changes on radiographs (Ahlbäck II- V).
* Malalignment on full-length radiographs showing increased stress in the involved knee compartment.
* Presence of associated ipsilateral ankle joint problem.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Lysholm knee score | baseline, 2 years postoperative
  functional knee score, minimum is zero, maximum value is 100, a higher score means a better outcome
Knee Injury and Osteoarthritis and Outcome (KOOS) score | baseline, and 2 years postoperative
  osteoarthritis knee score, minimum is zero, maximum is 100, higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H khalil, M.D, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronnblad E, Rotzius P, Eriksson K. Autologous semitendinosus tendon graft could function as a meniscal transplant. Knee Surg Sports Traumatol Arthrosc. 2022 May;30(5):1520-1526. doi: 10.1007/s00167-021-06606-8. Epub 2021 Jun 8. PMID 34100999
- [Background] Kohn D. Autograft meniscus replacement: experimental and clinical results. Knee Surg Sports Traumatol Arthrosc. 1993;1(2):123-5. doi: 10.1007/BF01565466. PMID 8536007
- [Background] Johnson LL, Feagin JA Jr. Autogenous tendon graft substitution for absent knee joint meniscus: a pilot study. Arthroscopy. 2000 Mar;16(2):191-6. doi: 10.1016/s0749-8063(00)90035-5. PMID 10705332
- [Background] Milenin O, Strafun S, Sergienko R, Baranov K. Lateral Meniscus Replacement Using Peroneus Longus Tendon Autograft. Arthrosc Tech. 2020 Jul 22;9(8):e1163-e1169. doi: 10.1016/j.eats.2020.04.016. eCollection 2020 Aug. PMID 32874897